CLINICAL TRIAL: NCT06820580
Title: The Effect of Salutogenic Approach Based Interview on Subjective Recovery and Quality of Life in Individuals With Schizophrenia
Brief Title: The Effect of Salutogenic-based Interviewing on Subjective Recovery and Quality of Life in Schizophrenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Şeyda Erçel, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU-SBF-ŞE-01
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Salutogenesis; Subjective Recovery; Quality of Life
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: A randomized controlled study design will be used. It is planned to include 30 individuals in the experimental group and 30 individuals in the control group by randomization method (using the software at http://www.randomizer.org). Participants will be divided into two groups:
  Experimental group Control group Individuals in the experimental group will be subjected to a four-week training program and assessments will be made twice, before and after the training. In the control group, no training will be given and the assessments will be conducted twice, four weeks apart.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salutogenic Approach Based Interview Group (Experimental): Participants will be offered an 8-session Salutogenic Approach Based Interview Program two days a week.
  Interventions: Other: Salutogenic Approach Based Interview
- Control group (No Intervention): There will be no intervention interview. They will continue their normal routines and treatments at the community mental health center.

INTERVENTIONS:
Other: Salutogenic Approach Based Interview — Salutogenic Approach Based Interviewing Program consists of 8 sessions. The interview will be conducted for four weeks and on two specific days of the week. Interviews will be conducted in groups of 6-8 people. The interview will last 30-40 minutes on average.
  Arms: Salutogenic Approach Based Interview Group

SUMMARY:
Schizophrenia is an inherited, complex, multidimensional syndrome with varying degrees of psychotic, negative, cognitive, mood and motor symptoms. Schizophrenia is a serious public health problem that causes significant losses in the lives of individuals due to both its occurrence at a young age and its prevalence. Ranked by the World Health Organization as one of the top ten diseases contributing to the global burden of disease, it is among the most disabling and economically disastrous medical disorders. The boundaries of schizophrenia remain unclear, indicating a lack of categorical cohesion and the need to reconceptualize it as a broader, multidimensional and/or spectrum construct.

With the discovery of antipsychotic drugs, the symptoms of the disease were alleviated, the level of severity decreased and the length of hospitalization was shortened. However, this led to repeated hospitalizations of patients with chronic course and a revolving door effect occurred. Drug treatment has a limited effect on readjustment to society, improving social relations and increasing self-care activities in individuals with chronic mental illness. Therefore, it is important to support drug treatment with social support programs and various psychosocial approaches. In the past, pathogenic approaches focusing on problems and risk factors have been adopted to promote and maintain health. The salutogenic model developed by medical sociologist Aaron Antonovsky (1987) focuses on the causes of health rather than the factors that cause disease. This model is concerned with the relationship between how people approach stressful situations (such as mental and chronic health conditions and their consequences) and their individual ability to self-manage and cope with these situations. The model is a medical approach that focuses on the causes of health rather than the factors that cause disease.

This study was planned to evaluate the effect of salutogenic approach-based interviewing on subjective recovery and quality of life in individuals diagnosed with schizophrenia.

DETAILED DESCRIPTION:
Salutogenesis theory focuses on what contributes to the development of good health and contrasts with pathogenesis explaining disease. The most important question for the salutogenic orientation is how a person identifies and utilizes different resources and thus how health promotion can be supported. It focuses on the creation and maintenance of good health rather than looking for the cause of specific diseases. This is in contrast to the traditional pathogenic model, which focuses on risk factors that play a role in disease occurrence.

The similarity between the core principle of the salutogenic model and the professional purpose of psychiatric nursing is striking. Psychiatric nursing supports the protection and promotion of community mental health, the rehabilitation of disorders and the regaining of the ability to cope with the experiences of suffering and to find meaning in life. Therefore, the model is suitable for many practice areas of psychiatric nurses.

The increasing number of people living with mental health problems in society for many years focuses on the need for recovery from a coping and mental health promotion perspective. The value of salutogenic theory is that it emphasizes coping and health promotion. Although there are numerous empirical applications of salutogenic theory in the field of public health, reviews of salutogenic-based interventions and their impact on population health are limited. Through the salutogenic method, examining deep challenges can provide opportunities to understand how individuals cope during crises and suggest methods to improve the health of the general population. As nursing education and intervention, it is important in terms of emphasizing the need for health promotion and ultimately promoting normal physical and psychological health.

The motto of the Mental Health Action Plan for 2021-2023 is stated as "Implementing an integrated community-based mental health service model in mental health services, monitoring, protecting and improving the mental health of individuals". Subjective recovery is a personally perceived improvement that includes other factors beyond clinical recovery. These factors focus on areas of personal development such as empowerment, having a sense of hope, having confidence in the future, redefining oneself, overcoming stigmatization, establishing supportive relationships, taking responsibility, giving meaning to life and leading a fulfilling life. Subjective well-being and quality of life are increasingly recognized as important treatment outcomes in patients with schizophrenia. Schizophrenia, which usually lasts a lifetime, is a disorder that causes significant problems in quality of life and functioning. Factors such as physical health, adaptability, well-being, economic status and social interaction are among the components of quality of life.

Therefore, this study was planned to evaluate the effect of salutogenic approach-based interviewing on subjective recovery and quality of life in individuals diagnosed with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* The participant is in the recovery (remission) period
* Being diagnosed with schizophrenia
* Being suitable for group work

Exclusion Criteria:

* The participant experienced an exacerbation (relapse) period
* Presence of hearing and comprehension problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-10-26 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Subjective Recovery Assessment Scale | From immediately before the interview began to 4 weeks after the interview.
  It is a 17-item Likert-type self-report scale. Each item is scored from 1 to 5. Higher scores indicate that the individual perceives himself/herself as more recovered. The scale has no sub-dimensions and is evaluated as a single factor. Cronbach's alpha coefficient of the scale was found to be 0.987.

SECONDARY OUTCOMES:
Quality of Life Scale for Schizophrenia | From immediately before the interview began to 4 weeks after the interview.
  The scale, which is administered in a semi-structured interview and assessed by the interviewer, is designed to assess the quality of life of schizophrenia patients receiving maintenance treatment. The scale provides information about symptoms and functioning over the previous four weeks. It consists of 21 questions and four sub-dimensions: interpersonal relationships (questions 1-8), occupational role (questions 9-12), mental symptoms (questions 13-17 and 20-21), and daily use and activities (questions 18-19). Each item consists of three parts. In the first part, a brief description is given to help the interviewer understand and focus on the parameter to be assessed, in the second part, a few sample questions are given to help the interviewer examine the patient, and in the third part, a 7-point Likert-type scale is given to make the assessment. The Cronbach Alpha reliability coefficient of the scale was found to be 0.80.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda Erçel, MSc, Principal Investigator — Ataturk University; Sibel Asi Karakaş, Principal Investigator — Ataturk University
Locations (1):
- Elazığ Community Mental Health Center, Elâzığ, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No